CLINICAL TRIAL: NCT01839175
Title: A Phase III Open-label Randomised Study to Evaluate the Immunogenicity and Safety of the Concomitant Administration of a New Hexavalent DTaP-IPV-HepB-PRP-T Combined Vaccine (Hexavalent Vaccine) Given at 2, 3, and 4 Months of Age With a Meningococcal Serogroup C Conjugate (MenC) Vaccine Given at 2 and 4 Months of Age
Brief Title: Concomitant Administration of a New Hexavalent Vaccine With a Meningococcal Serogroup C Conjugate Vaccine in Healthy Infants During Primary Series Immunisation Followed by Booster Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HXM01C; 2012-005547-24 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Neisseria Meningitidis; Bacterial Infections; Virus Diseases
MeSH Terms: conditions — Bacterial Infections; Virus Diseases | interventions — Vaccines, Combined; Tetanus Toxoid; Hepatitis B Vaccines; 13-valent pneumococcal vaccine; Pneumococcal Vaccines; RotaTeq; Vaccines; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: Hexavalent vaccine; Biological: NeisVac-C; Biological: Prevenar 13; Biological: RotaTeq; Biological: Nimenrix; Biological: M-M-RVAXPRO
- Group 2 (Active Comparator)
  Interventions: Biological: Hexavalent vaccine; Biological: Prevenar 13; Biological: RotaTeq; Biological: Nimenrix; Biological: M-M-RVAXPRO

INTERVENTIONS:
Biological: Hexavalent vaccine — 0.5 mL intramuscular injection at 2, 3 and 4 months of age (primary series) 0.5 mL intramuscular injection at 12 or 13 months of age (booster)
  Other Names: Diphtheria, tetanus, pertussis, hepatitis B,; poliomyelitis and Haemophilus influenzae type b conjugate vaccine (adsorbed).
Biological: NeisVac-C — 0.5 mL intramuscular injection at 2 and 4 months of age
  Other Names: Meningococcal group C polysaccharide conjugate vaccine adsorbed
  Arms: Group 1
Biological: Prevenar 13 — 0.5 mL intramuscular injection at 2 and 4 months of age (primary series) 0.5 mL intramuscular injection at 13 months of age (booster)
  Other Names: Pneumococcal conjugate vaccine (13-valent, adsorbed)
Biological: RotaTeq — 2 mL oral administration at 2, 3 and 4 months
  Other Names: Human-bovine rotavirus reassortants (live) vaccine
Biological: Nimenrix — 0.5 mL intramuscular injection at 12 months
  Other Names: Meningococcal group A, C, W-135 and Y conjugate vaccine
Biological: M-M-RVAXPRO — 0.5 mL intramuscular or subcutaneous injection at 13 months of age
  Other Names: Measles, mumps and rubella vaccine (live)

SUMMARY:
Primary Series Primary objectives

* To demonstrate that the concomitant administration of the hexavalent vaccine with a meningococcal serogroup C conjugate vaccine is non inferior to the administration of the hexavalent vaccine without a MenC vaccine concomitantly in term of seroprotection rate for hepatitis B one month after the third dose of the hexavalent vaccine
* To demonstrate that the concomitant administration of a MenC vaccine with the hexavalent vaccine induces an acceptable response for MenC in term of seroprotection rate (SPR) one month after the second dose of MenC

Booster Primary objectives

- To describe the immunogenicity of a booster dose of the hexavalent vaccine and of a meningococcal group ACWY conjugate (MenACWY) vaccine either co-administered at 12 months of age or given separately.

DETAILED DESCRIPTION:
Primary Series Secondary objectives

* To describe the antibody response to all the hexavalent vaccine antigens one month after the third dose of the hexavalent vaccine when given concomitantly or not to MenC
* To describe the antibody response to MenC vaccine when a MenC vaccine is given concomitantly with the hexavalent vaccine, one month after the first and the second dose of MenC vaccine
* To describe the safety profile of the hexavalent vaccine after each and any injection when given concomitantly or not with a MenC vaccine

Booster Secondary objectives

* To describe the antibody (Ab) persistence at 12 months of age for the hexavalent valences following a 3-dose primary vaccination at 2, 3 and 4 months of age (prior to administration of a booster dose)
* To describe the safety of a booster dose of the hexavalent vaccine and of a meningococcal group ACWY conjugate (MenACWY) vaccine either co-administered at 12 months of age or given separately.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant 46 to 74 days of age (both inclusive)
* Born at full term of pregnancy (≥37 weeks) and/or with a birth weight≥2.5 kg
* Subject's parent(s) or legal representative able to comply with the study procedures

Exclusion Criteria:

* Participation in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding each study vaccination
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, poliomyelitis, Haemophilus influenzae type b, meningococcal, pneumococcal, rotavirus infection
* Know or suspected congenital, hereditary or acquired immunodeficiency
* History of seizures or encephalopathy
* Known thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection
* Chronic illness that could interfere with trial conduct or completion
* Known or suspected hypersensitivity to any of the study vaccines' active substance or excipients or history of a life-threatening reaction to a vaccine(s) containing the same substances as the study vaccines
* Contraindication to any of the study vaccines
* Known personal or maternal history of hepatitis B or hepatitis C seropositivity
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, Haemophilus influenzae type b or meningococcal serogroup C infection
* Receipt of immune globulin, blood or blood-derived products, immunosuppressive drugs, systemic corticosteroid since birth
* Identified as a natural or adopted child of the investigator or employee with direct involvement in the current study.

Ages: 46 Days to 76 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an anti-hepatitis B concentration ≥10 IU/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine)
Proportion of subjects with an anti-MenC titre ≥1:8 dil | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine)

SECONDARY OUTCOMES:
Proportion of subjects with an anti-polyribosylribitol phosphate concentration ≥0.15 µg/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with an anti-diphtheria concentration ≥0.01 IU/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster)
Proportion of subjects with an anti-tetanus concentration ≥0.01 IU/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster)
Proportion of subjects with an anti-inactivated poliovirus 1, 2, 3 titre ≥1:8 dil | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with pertussis vaccine response | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine)
Proportion of subjects with an anti-MenC titre ≥1:8 dil | Month 3 (One month after dose 1 of MenC vaccine)
Solicited injection-site and systemic reactions | Day 1 to Day 7 following vaccination
Unsolicited adverse events | Day 1 to Day 30 following vaccination
Serious adverse events | From signature of the informed consent to the last visit of the subject, an expected average of 11 months
Proportion of subjects with an anti-polyribosylribitol phosphate concentration ≥1 µg/mL | Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with an anti-diphtheria concentration ≥0.1 IU/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with an anti-tetanus concentration ≥0.1 IU/mL | Month 5 (One month after dose 3 of the hexavalent vaccine and dose 2 of MenC vaccine), Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with an anti-MenA, anti-MenC, anti-MenW-135, anti-MenY titre ≥1:8 dil | Month 13 (One month after MenAWCY vaccine)
Proportion of subjects with an anti-hepatitis B concentration ≥10 IU/mL | Month 12 (Pre-booster) and Month 13 (One month post-booster)
Proportion of subjects with pertussis booster response | Month 13 (One month post-booster)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (11):
- Finland (11):
  - Sanofi Pasteur MSD Investigational Site 003, Espoo
  - Sanofi Pasteur MSD Investigational Site 001, Helsinki
  - Sanofi Pasteur MSD Investigational Site 002, Helsinki
  - Sanofi Pasteur MSD Investigational Site 011, Jarvenpaa
  - Sanofi Pasteur MSD Investigational Site 010, Kokkola
  - Sanofi Pasteur MSD Investigational Site 004, Oulu
  - Sanofi Pasteur MSD Investigational Site 005, Pori
  - Sanofi Pasteur MSD Investigational Site 009, Seinäjoki
  - Sanofi Pasteur MSD Investigational Site 006, Tampere
  - Sanofi Pasteur MSD Investigational Site 007, Turku
  - Sanofi Pasteur MSD Investigational Site 008, Vantaa

REFERENCES:
- [Derived] Vesikari T, Borrow R, Da Costa X, Thomas S, Eymin C, Boisnard F, Lockhart S. Concomitant administration of a fully liquid ready-to-use DTaP-IPV-HB-PRP-T hexavalent vaccine with a meningococcal ACWY conjugate vaccine in toddlers. Vaccine. 2018 Dec 18;36(52):8019-8027. doi: 10.1016/j.vaccine.2018.10.100. Epub 2018 Nov 22. PMID 30471953
- [Derived] Vesikari T, Borrow R, Da Costa X, Richard P, Eymin C, Boisnard F, Lockhart S. Concomitant administration of a fully liquid, ready-to-use DTaP-IPV-HB-PRP-T hexavalent vaccine with a meningococcal serogroup C conjugate vaccine in infants. Vaccine. 2017 Jan 11;35(3):452-458. doi: 10.1016/j.vaccine.2016.11.053. Epub 2016 Dec 9. PMID 27939054